CLINICAL TRIAL: NCT04220034
Title: Autoantibodies Prevalence and Their Related-diseases During Checkpoint Inhibitor Treatment
Brief Title: Autoantibodies Prevalence During Checkpoint Inhibitor Treatment
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA19123*
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Autoimmune Adverse Effects of Anti-neoplasic Drug
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients receiving inhibitor checkpoint treatment: adult patients that will receive for the first time checkpoint inhibitor for a neoplasic disease in a center participating to the study
  Interventions: Biological: Blood sample

INTERVENTIONS:
Biological: Blood sample — Blood sample will be collected to determine development or increase level frequencies of different types of autoantibodies in patients receiving ICI for the first time

SUMMARY:
The use of Checkpoint inhibitors (ICIs) is rapidly expanding to the treatment of many cancer types. Autoimmunity and clinical autoimmune diseases represent adverse events of ICIs with variable severity and consequences. Clinical trials using ICIs have largely excluded patients with preexisting autoimmune diseases but the rate of autoimmune flares has been reported to be high in patients with preexisting autoimmune diseases in retrospective cohort studies. Moreover numerous retrospective cases and series reported ICI-related autoimmune diseases in patients without any previous autoimmune event.

To date, no study has prospectively evaluated the rate of biological and clinical autoimmunity in patients. Moreover, guidelines concerning autoantibodies monitoring in patients are subject of debate.

DETAILED DESCRIPTION:
The aim of this prospective study is to determine development or increase level frequencies of different types of autoantibodies in patients receiving ICI for the first time. The rate of clinical autoimmunes diseases development will also be recorded and correlated with autoantibodies prevalence before and during ICI treatment.

Results will help to determine the rate of biological and clinical autoimmune events induced by ICIs in unselected patients and will help to clarify autoimmunity screening strategy in this setting.

ELIGIBILITY:
Inclusion Criteria:

* patients receiving check point inhibitor for a neoplasic disease in a center that participates to the study during the inclusion period
* patients who agree to participate in the study
* adult patients (aged more than 18 years old)

Exclusion Criteria:

- previous treatment with check point inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving inhibitor checkpoint treatment
Sampling Method: Non-Probability Sample
Enrollment: 183 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
development or increase level of anti-nuclear antibody | Month 6
  Development of anti-nuclear antibody will be defined by detection of autoantibodies above the positive threshold of the test if below the positive threshold initially (seroconversion) Increase level of anti-nuclear antibody will be defined by increase of at least 2 dilutions of the antibody titer
development or increase level of anti-cyclic citrullinated peptide antibodies | Month 6
  Development of anti-cyclic citrullinated peptide antibodies will be defined by detection of autoantibodies above the positive threshold of the test if below the positive threshold initially (seroconversion) Increase level of anti-cyclic citrullinated peptide antibodies will be defined by doubling the concentration of the antibody titer
development or increase level of rheumatoid factor | Month 6
  Development of rheumatoid factor will be defined by detection of autoantibodies above the positive threshold of the test if below the positive threshold initially (seroconversion) Increase level of rheumatoid factor will be defined by doubling the concentration of the antibody titer
development or increase level of Anti-glutamic acid decarboxylase antibodies | Month 6
  Development of Anti-glutamic acid decarboxylase antibodies will be defined by detection of autoantibodies above the positive threshold of the test if below the positive threshold initially (seroconversion) Increase level of Anti-glutamic acid decarboxylase antibodies will be defined by doubling the concentration of the antibody titer
development or increase level of Anti-thyroperoxydase antibodies | Month 6
  Development of anti-TSH receptor antibodies will be defined by detection of autoantibodies above the positive threshold of the test if below the positive threshold initially (seroconversion) Increase level of anti-TSH receptor antibodies will be defined by doubling the concentration of the antibody titer
development or increase level of Auto-antibodies associated with myositis | Month 6
  Development of Auto-antibodies associated with myositis antibodies will be defined by detection of autoantibodies above the positive threshold of the test if below the positive threshold initially (seroconversion) Increase level of Auto-antibodies associated with myositis antibodies will be defined by doubling the concentration of the antibody titer

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided